CLINICAL TRIAL: NCT03773120
Title: Effectiveness of Intraoperative Neuromonitoring of the External Branch of the Superior Laryngeal Nerve During Thyroid Surgery
Brief Title: Effectiveness of Intraoperative Neuromonitoring of External Branch of Superior Laryngeal Nerve During Thyroid Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Major study protocol changes
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Su-jin Kim, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1708-125-880
Record Dates: First submitted 2018-04-12; First posted 2018-12-12 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Carcinoma, Papillary, Follicular
Keywords: superior laryngeal nerve
MeSH Terms: conditions — Carcinoma, Papillary, Follicular

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using Neuromonitoring to find EBSLN (Experimental): With Neuromonitoring of the EBSLN using nerve monitoring system
  Interventions: Device: Using Neuromonitoring to find EBSLN
- No Using Neuromonitoring to find EBSLN (No Intervention): Without Neuromonitoring of the EBSLN using nerve monitoring system

INTERVENTIONS:
Device: Using Neuromonitoring to find EBSLN — intraoperative neuromonitoring to preserving external branch of superior laryngeal nerve during thyroid surgery
  Arms: Using Neuromonitoring to find EBSLN

SUMMARY:
The paralysis of the external branch of superior laryngeal nerves after thyroid surgery is known to be a common complication resulting in poor quality of life. Aim of this randomized control trial(RCT) is to evaluate effectiveness of neuromonitoring during thyroid surgery for the preservation of these nerves.

DETAILED DESCRIPTION:
The external branch of superior laryngeal nerves(EBSLNs) are important for voice quality. Injury to this nerve during thyroid surgery can manifest as ipsilateral paralysis of the cricothyroid muscle. Clinical symptoms may include: hoarseness, breathy voice, an increase in the rate of throat clearing, vocal fatigue, or diminished vocal frequency range, especially with regards to raising pitch. The amount of EBSLNs identified intraoperatively varies from 10% to 80%, while the rate of EBSLN injury reported in the literature is between 5% and 28%, depending on different evaluation methods. Advances in intraoperative neuromonitoring techniques would allow for EBSLN identification during thyroid surgery. However, there is controversy regarding usefulness in preserving EBSLN function using nerve monitoring system. The aim of the study is to evaluate effectiveness of neuromonitoring during thyroid surgery for the preservation of EBSLNs.

ELIGIBILITY:
Inclusion Criteria:

* planned open thyroidectomy
* acceptable clinical laboratory tests
* understand clinical trials
* no significant past medical history

Exclusion Criteria:

* planned radical neck dissection
* hyperthyroidism history
* history of laryngeal nerve palsy
* laryngeal disease history
* uncontrolled hypertension or diabetes mellitus or heart disease
* anticoagulation or antiplatelet medication
* stroke history
* participated another clinical trials in 30days

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Identification of EBSLN during thyroid surgery | up to postoperative 12 months
  Identification rate of EBSLN

SECONDARY OUTCOMES:
Location of EBSLN | up to postoperative 12 months
  Classification of EBSLN according to Cernea classification
Vocal outcome | up to postoperative 12 months
  Voice assessment using voice lab

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided